CLINICAL TRIAL: NCT06867159
Title: Comparison of Effects of Autogenic Inhibition and Reciprocal Inhibition Muscle Energy Techniques on Iliotibial Band Syndrome
Brief Title: Autogenic Inhibition Versus Reciprocal Inhibition Muscle Energy Techniques in Iliotibial Band Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FUI/CTR/2025/3
Record Dates: First submitted 2025-03-04; First posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Iliotibial Band Syndrome
MeSH Terms: conditions — Iliotibial Band Syndrome

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Outcomes Assessor
Masking Description: It will be a single blinded RCT in which assessor will be blinded to the group allocation of participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Autogenic Inhibition (AI) MET Group (Experimental): Autogenic Inhibition (AI) MET (Post Facilitation Stretch)
  1. The shortened muscle (Tensor Fascia Latae) is placed in a mid-range position about halfway between a fully stretched and a fully relaxed state.
  2. The patient contracts the muscle isometrically, using a maximum degree of effort for 5-10 seconds while the effort is resisted completely.
  3. On release of the effort, a rapid stretch is made to a new barrier, without any 'bounce', and this is held for at least 10 seconds.
  4. The patient relaxes for approximately 20 seconds and the procedure is repeated between three and five times more.
  Interventions: Procedure: Autogenic Inhibition (AI) MET (Post Facilitation Stretch)
- Reciprocal Inhibition (RI) MET Group (Experimental): Reciprocal Inhibition (RI) MET
  1. The shortened muscle (Tensor Fascia Latae) is placed in a mid-range position about halfway between a fully stretched and a fully relaxed state.
  2. The patient contracts the antagonist muscles (hip adductors), using a maximum degree of effort for 5-10 seconds while the effort is resisted completely.
  3. On release of the effort, a rapid stretch to TFL is made to a new barrier, without any 'bounce', and this is held for at least 10 seconds.
  4. The patient relaxes for approximately 20 seconds and the procedure is repeated between three and five times more.
  Interventions: Procedure: Reciprocal Inhibition (RI) MET

INTERVENTIONS:
Procedure: Autogenic Inhibition (AI) MET (Post Facilitation Stretch) — Autogenic Inhibition (AI) MET (Post Facilitation Stretch)
  1. The shortened muscle (Tensor Fascia Latae) is placed in a mid-range position about halfway between a fully stretched and a fully relaxed state.
  2. The patient contracts the muscle isometrically, using a maximum degree of effort for 5-10 seconds while the effort is resisted completely.
  3. On release of the effort, a rapid stretch is made to a new barrier, without any 'bounce', and this is held for at least 10 seconds.
  4. The patient relaxes for approximately 20 seconds and the procedure is repeated between three and five times more.
  Arms: Autogenic Inhibition (AI) MET Group
Procedure: Reciprocal Inhibition (RI) MET — Reciprocal Inhibition (RI) MET
  1. The shortened muscle (Tensor Fascia Latae) is placed in a mid-range position about halfway between a fully stretched and a fully relaxed state.
  2. The patient contracts the antagonist muscles (hip adductors), using a maximum degree of effort for 5-10 seconds while the effort is resisted completely.
  3. On release of the effort, a rapid stretch to TFL is made to a new barrier, without any 'bounce', and this is held for at least 10 seconds.
  4. The patient relaxes for approximately 20 seconds and the procedure is repeated between three and five times more.
  Arms: Reciprocal Inhibition (RI) MET Group

SUMMARY:
Comparison of effects of autogenic inhibition and reciprocal inhibition muscle energy techniques on iliotibial band syndrome

DETAILED DESCRIPTION:
A single-blinded randomized control trial will be conducted over a period of one year in Foundation University Islamabad. Forty participants will be assigned to two groups: Group A (AI) and Group B (RI), with 20 participants each. The AI technique will involve a maximal isometric contraction of the target muscle followed by a stretch, while the RI technique will involve a maximal isometric contraction of the antagonist muscle followed by a similar stretching protocol. Both groups will perform the exercises 3 times per week for 2 weeks. Pain, Hip range of motion (ROM) and lower extremity function will be assessed using Numeric Pain Rating Scale (NPRS), goniometer and Lower Extremity Functional Scale (LEFS) respectively.

The outcomes will be measured in terms of improvements in pain score (NPRS), hip range of motion (ROM), and overall lower extremity function.

ELIGIBILITY:
Inclusion Criteria

* Both male and female participants
* Age : 19-45years (8)
* Lateral knee pain (>3 months)
* Tenderness over lateral femoral condyle
* Positive Flexibility Tests
* Modified Ober's test (9)
* Length assessment of Tensor Fasciae Latae and Iliotibial Band (10)
* Positive Pain Provocation Tests
* Renne's test
* Noble's Compression test (11) *(individuals with 3 positive tests out of above mentioned 4 tests will be included)

Exclusion Criteria

* Recent lower limb or pelvic girdle surgery within the past 3 months
* Lower limb fractures or trauma within the past year.
* Multiple lower limb surgeries (>2)
* Presence of any structural or postural disorders (kyphosis or severe scoliosis)
* Neurological disorders
* Hip and knee Osteoarthritis
* Rheumatoid Arthritis
* Pregnancy

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-07-15 (Estimated)

PRIMARY OUTCOMES:
Pain severity | 2 weeks
  Pain will be assessed using Numeric Pain Rating Scale (NPRS),
Range of motion | 2 weeks
  Hip range of motion (ROM) will be assessed using goniometer
Functional status of lower limb | 2 weeks
  Lower extremity function will be assessed using Lower Extremity Functional Scale (LEFS)

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physcial Therapy, Rawalpindi, Punjab Province, Pakistan